CLINICAL TRIAL: NCT04272164
Title: Effects of Weighted Rope Jump Training on Physical Fitness in Taekwando Athletes
Brief Title: Weighted Rope Training in Taekwando Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Fatima iftikhar REC-0577
Record Dates: First submitted 2020-02-13; First posted 2020-02-17 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Physical Performance
Keywords: Taekwondo; Physical fitness,; weighted rope jump training.

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- technical taekwondo training (Active Comparator): Light jogging,running, Stretching exercises,Pushups and sit ups, Punches,Kicks
  Interventions: Other: technical taekwando training
- weighted rope taekwondo training (Experimental): weighted rope jump training along with tachnical taekwando training
  Interventions: Other: technical taekwando training; Other: weighted rope jump training

INTERVENTIONS:
Other: technical taekwando training — Light jogging followed by star jump, Different running styles (forward, backward and sideways), Stretching exercises (Upper and lower Limb), Pushups and sit ups, Punches (single, double, triple, nonstop punches including speed and power, punches with forward and backward stepping), Kicks (rising kick, front kick, middle kick, drop kick ( in +out+center), Stances (walk stance, punching stance, front deep stance, kicking stance), Blockings (solar block, upper block and lower block), Self -defense (neck gripping, hand gripping, locking), Sand bag drills, Balance training 10 repeatitions of 1 set each, 3 days a week for 8 weeks
Other: weighted rope jump training — Basic bounce step with both feet 2. Bell jump with both feet 3. Skier's jump 4. Right foot skipping 5. Left foot skipping, 6. Alternate foot step 7. Boxer shuffle 8. Side straddle 9. Scissors 10. Bonus jump with both feet After the preparatory weighted rope jump training (WRJT) for 1 week, subjects in experimental group followed jumping training by repetition method 3 days in a week for 8 weeks in addition to the routine taekwondo training program. 3 sets per week with 30 seconds training duration and 30 seconds rest duration. with progressive increase in the intensity and no. of sets.
  Arms: weighted rope taekwondo training

SUMMARY:
The aim of this study was to determine the effects of weighted rope jump training on physical fitness in taekwondo athletes. Randomized controlled trail was done on Total 52 male taekwondo players, aged between 13 to 19 years. Players were randomly divided into 2 groups at Khubaib Taekwondo Academy. Experimental group ( n=26) had weighted rope training for 8 weeks, 3 days in a week along with routine taekwondo training and control group (n=26) had to follow only routine training for 8 weeks. Agility t- test, 50 meter run test, sargent jump test, sit and reach test and yo-yo endurance test were performed at baseline, 4th and 8th week to assess the physical fitness in participants. Hand grip dynamometer was used to assess the upper limb strength.

DETAILED DESCRIPTION:
Taekwondo (TKD) means "fight with foot and fist" is a very energetic, quick sport. Kicks and punches are used with full force by the athletes to knock down their opponents. Taekwondo (TKD) is one of the most systematic traditional combat practice and fighting sports in Korea that has high status in the world. Taekwondo originated from Korea and has been playing as an Olympic sports since 2000. Presently, it is practiced in 2 methods under International Taekwondo Federation (ITF) and World Taekwondo Federation (WTF). Games are organized on the basis of age, weight, height and gender at national and international level.

In beginning, basic skills are taught to athletes which consist of strikes, blocks, kicking techniques, stances and different form. Taekwondo (TKD) is recognized by using very fast and high kicks. For this, athletes should be physically fit and active. Muscle strength, power, endurance, flexibility, agility, speed and cardiopulmonary endurance are the main components of physical fitness. Ability of muscle to generate maximum pressure voluntarily is called muscle strength. The force generated in a particular motion is called power. Capability of muscle to produce force against maximal resistance is known as endurance. Agility is ability to change direction while maintaining body balance. Speed is described as the shortest time requisite for an object to travel along a fixed distance. Flexibility is defined as an ability of a joint to move freely. In taekwondo sports both aerobic and anaerobic fitness are required but anaerobic energy contributes a lot during the fight.

Taekwondo is a contact sport and as compared to other martial arts, rate of injuries in taekwondo is very high. During kick, the knee is always in extended position. Quadriceps, hamstrings and calf muscles are activated at different times. Gluteal work as stabilizers during kick. Injuries may occur during fight (54%) as well as during training (36%). Lower limb injuries most common (46%) and upper limb injuries are (18%). Less injuries occur in vertebral areas (10%) and skull area (3%). Agility, flexibility, reactivity, endurance, strength and speed are the main factors related to physical fitness and are important in taekwondo (TKD).

Rope jumping training is very effective in improving muscle work, physical fitness and cardiorespiratory endurance. For many sports activities along with kick boxing, fighting, badminton, and combat sports, skipping rope training is a major training tool. Along with rope jump training, weighted rope jumping protocol has also gain importance in improving physical fitness and athletes' performance. Weighted ropes are made up of hard plastic or steel material having different weights in handle and rope portion. Weighted ropes are usually utilized in 2 specific ways. If weight is only present in handles then its mean it will improve lower limb strength, coordination, speed, response and flexibility. If weight is present in both handles and rope portion, the training will show better results for both upper and lower limb strength and coordination. So, in most of the trainings, weighted rope jumping (WRJ) is recommended in order to achieve its useful effects for both upper limb and lower limb.

In 2018, conducted a research work to see the effects of neuromuscular weighted rope jumping training on lower extremity reaction time. Pre and post training visual and auditory response time of both dominant and non-dominant leg was assessed by Opto Jump System and the result indicated that the weighted rope training program is effective in decreasing the reaction time.

In 2017, investigated the effect of simple rope jumping and weighted rope jumping exercise protocol on body structure and strength performance of young women volleyball athletes. The result showed significant improvement in strength and endurance of both upper and lower limb in weighted rope training group.

In 2016, compared the effects of 12-week normal rope jumping protocol with weighted rope jumping training on physical health assessments along with anaerobic efficency, speed, agility and flexibility in girls adolescent volleyball athletes and in the end anaerobic fitness and agility was significantly improved in experimental group.

In 2011 conducted a study to know the outcomes of simple rope skipping or weighted rope skipping training on strength, coordination and proprioception in girls volleyball participants in which results showed that the weighted rope jump protocol group was the most improved group.

In 2015, Speed and Jumping-rope training protocol on fine motor skills of female school population.SO, it was suggested that rope skipping method can be used as a right program for the development of fine motor skills.

In 2013, the study done, it aim to analyze results of weighted rope jumping training (WRJT) performed by repetition procedure on physical fitness and response time of basketball athletes and weighted rope had improved results of heart rate and anaerobic fitness.

ELIGIBILITY:
Inclusion Criteria:

* Male taekwondo players .

  * Athletes having experience of minimum one year
  * Athletes already following taekwondo training program
  * Participants falling in Bantam to light middle weight category

Exclusion Criteria:

* • Having had upper and lower extremity pain in movement rated at least 3/10 on Numeric Pain Rating scale.

  * Having a systemic pathology including inflammatory joint disease.
  * Having had active intervention related to upper or lower extremity pathology in last 3 months
  * Having taken anti-inflammatory medication in the past two weeks.

Ages: 13 Years to 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 52 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
digital Hand grip dynamometer | 8 week
  Handgrip Dynamometers are instruments for measuring the maximum isometric strength of the hand and forearm muscles, used for testing handgrip strength of athletes involved in strength training. the person applies maximum force on the dynamometer by griping. the reading is noted for both right and left hand.

SECONDARY OUTCOMES:
agility T-test | 8 week
  Purpose of agility t- test was to see directional changes in athletes and includes forward, lateral, and backwards running. 3 cones were arranged in the shape of T. Starting point of test was A and ending point was also A. Distance between cone A and B was 10 yards and distance between cone B to C and B to D was 5 yards As the stop watch started, the player started running from point A to point B and touched the cone with right hand. Then started sideways running from cone B to cone C and touched the cone with left hand and again sideways running from cone C to D and touched the cone D with right hand.
  Males (seconds) Females (seconds) Excellent < 9.5 < 10.5 Good 9.5 to 10.5 10.5 to 11.5 Average 10.5 to 11.5 11.5 to 12.5 Poor > 11.5 > 12.5 Again coming back to cone B touching it with left hand, player started backward running towards cone A. This is the finishing line of T- test. This test was performed 3 times and average score was recorded in seconds.
50 meter sprint test | 8 week
  Purpose of sprint test was to check speed and acceleration of athlete. In this test, 50 meter distance was measured by measuring tape. Cone A was placed at starting point A and cone B at the finishing point. As the timer started, player started running with speed from cone A to cone B. This test was performed 3 times and the average score was recorded in seconds.
Sargent jump test | 8 week
  The aim of sargent jump test was to assess the strength of lower limb. In this test we need a measuring tape and a chalk. Player was instructed to stand with his right shoulder to the side of the wall and touched the wall with his right hand. This was his normal reach height that was point A. In second part of this test player was instructed to take high jump and touched the wall as far as his can reach. This was marked as B. In the end difference of point A and B was taken (B-A). Test readings were taken 3 times and the jumping height was documented in cm.
Sit and reach test | 8 week
  Sit and reach test was performed to know the flexibility of low back and hamstring muscles. In this test we need a box and a measuring tape. Player was instructed to sit on the floor with shoes removed, knees straight and feet touching the box. Instructions were given to bend forward and move the fingers on the box. Distance was measured from the tip of fingers to the edge of box. Test was performed 3 times and average score was recorded in cm
Yo Yo endurance test | 8 week
  The purpose of Yo-Yo endurance test was to evaluate the cardiorespiratory endurance (aerobic fitness). In this test we need 3 cones and audio of yo yo endurance test. Distance between cone A to cone B was 5meter which is the resting time for 10s. From cone B to C distance was 20 meter. Starting point of Test was cone B. As the audio started in 5 seconds with beep sound, players started running from point B to point C and back to point B without taking rest. From point B to A was recovery time for players and as the next beep sound heard, the test again started. This test consist of different levels and it depends on players' endurance that how effectively they can perform this test. Players can quit at any level if he got exhausted. Warnings are given if athletes do not reach the starting and finishing line with the sound of beep. Scores recorded as levels.

CONTACTS AND LOCATIONS:
Overall Officials: Aisha Razzaq, MS-OMPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah International university, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pingale N, Ghagare J. Prevalence of musculoskeletal injuries in young taekwondo athletes. 2017.
- [Background] Fong SS, Ng GY. Does Taekwondo training improve physical fitness? Phys Ther Sport. 2011 May;12(2):100-6. doi: 10.1016/j.ptsp.2010.07.001. PMID 21496773
- [Background] Lee SM, Ricke G. Official taekwondo training manual: Sterling Publishing Company, Inc.; 2005.
- [Background] Noorul H, Pieter W, Erie Z. Physical fitness of recreational adolescent taekwondo athletes. Brazilian Journal of Biomotricity. 2008;2(4):230-40.
- [Background] Santos VG, Franchini E, Lima-Silva AE. Relationship between attack and skipping in Taekwondo contests. J Strength Cond Res. 2011 Jun;25(6):1743-51. doi: 10.1519/JSC.0b013e3181ddfb0f. PMID 21512402
- [Background] Tornello F, Capranica L, Chiodo S, Minganti C, Tessitore A. Time-motion analysis of youth Olympic Taekwondo combats. J Strength Cond Res. 2013 Jan;27(1):223-8. doi: 10.1519/JSC.0b013e3182541edd. PMID 22592166
- [Background] Miller TA. National Strength and Conditioning Association (NSCA)'s Guide to Tests and Assessments. 2012.
- [Background] Chiodo S, Tessitore A, Cortis C, Lupo C, Ammendolia A, Iona T, Capranica L. Effects of official Taekwondo competitions on all-out performances of elite athletes. J Strength Cond Res. 2011 Feb;25(2):334-9. doi: 10.1519/JSC.0b013e3182027288. PMID 21233770
- [Background] Singh A, Boyat A, Sandhu J. Effect of a 6 week plyometric training pro-gram on agility, vertical jump height and peak torque ratio of Indian Tae-kwondo players. Sport Exerc Med Open J. 2015;1(2):42-6.
- [Background] Sheppard JM, Young WB. Agility literature review: classifications, training and testing. J Sports Sci. 2006 Sep;24(9):919-32. doi: 10.1080/02640410500457109. PMID 16882626
- [Background] Wasik J. Structure of movement of a turning technique used in the event of special techniques in Taekwon-do ITF. Archives of Budo. 2009;5:111-5.
- [Background] Turner AN. Strength & conditioning for Taekwondo athletes. Professional Strength & Conditioning. 2009(15):15-27.
- [Background] Fortina M, Mangano S, Carta S, Carulli C. Analysis of Injuries and Risk Factors in Taekwondo during the 2014 Italian University Championship. Joints. 2017 Aug 4;5(3):168-172. doi: 10.1055/s-0037-1605390. eCollection 2017 Sep. PMID 29270548
- [Background] Gleim GW, McHugh MP. Flexibility and its effects on sports injury and performance. Sports Med. 1997 Nov;24(5):289-99. doi: 10.2165/00007256-199724050-00001. PMID 9368275
- [Background] IPEKOGLU G, Erdogan CS, Er F, BALTACI G, COLAKOGLU FF. Effect of 12 week neuromuscular weighted rope jump training on lower extremity reaction time. world. 2018;8:5.
- [Background] Ozer D, Duzgun I, Baltaci G, Karacan S, Colakoglu F. The effects of rope or weighted rope jump training on strength, coordination and proprioception in adolescent female volleyball players. J Sports Med Phys Fitness. 2011 Jun;51(2):211-9. PMID 21681154
- [Background] Pulur A. The effects of weighted rope training on muscle damage of basketball players. International Journal of Physical Sciences. 2010;5(11):1787-95.
- [Background] Orhan S. Effect of weighted rope jumping training performed by repetition method on the heart rate, anaerobic power, agility and reaction time of basketball players. Advance in Environmental Biology. 2013;7:945-51.
- [Background] Turgut E, Çolakoğlu FF, Güzel NA, Karacan S, Baltacı G. Effects of Weighted Versus Standard Jump Rope Training on Physical Fitness in Adolescent Female Volleyball Players: A Randomized Controlled Trial. Fizyoterapi Rehabilitasyon. 2016;27(3):108-15.
- [Background] Lee B. Jump rope training: Human Kinetics; 2010.
- [Background] Khanjani M, Nourbakhsh P, Sepasi H. Effects of jumping-rope training on fine motor skills. Trends in Life Sciences. 2015;4(1):164-9.
- [Background] Duzgun I, Baltaci G, Colakoglu F, Tunay VB, Ozer D. The effects of jump-rope training on shoulder isokinetic strength in adolescent volleyball players. J Sport Rehabil. 2010 May;19(2):184-99. doi: 10.1123/jsr.19.2.184. PMID 20543219
- [Background] Partavi S. Effects of 7 weeks of rope-jump training on cardiovascular endurance, speed, and agility in middle school student boys. Sport Science. 2013;6(2):40-3.
- [Background] Haghighi AH, Cheraghian J, Hamedinia MR, Harati J. Comparing the Effect of a Jump Rope Training on Physical and Motor Fitness Components Among Primary School Boy and Girl Students.